CLINICAL TRIAL: NCT00897130
Title: Clinical and Biological Effects of 5-Azacitidine Five Days/Monthly Schedule in Symptomatic Low-risk Myelodysplastic Syndromes (MDSs)
Brief Title: 5-Azacitidine in Low-risk Myelodysplastic Syndromes (MDSs)
Acronym: MDSAZA0706
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Collaborators: University of Udine (Other); University of Bologna (Other); University of Genova (Other); University of Siena (Other); Cremona (Unknown); Mantova (Unknown)
Responsible Party: Principal Investigator, Domenico Russo, Full Professor of Hematology, Università degli Studi di Brescia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-003943-55
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Myelodysplastic Syndrome
Keywords: low-risk (IPSS 0-INT1) MDS according to WHO classification
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azacytidine (Experimental): Azacitidine will be given at a dose of 75mg/sqm subcutaneous daily for 5 consecutive days every 28 days (every month) for a total of 8 courses. 5-Aza dosages will be adjusted.
  Interventions: Drug: Azacytidine

INTERVENTIONS:
Drug: Azacytidine — Azacitidine will be given at a dose of 75mg/sqm subcutaneous daily for 5 consecutive days every 28 days (every month) for a total of 8 courses. 5-Aza dosages will be adjusted

SUMMARY:
Azacitidine will be given at a dose of 75 mg/sqm (s.c) daily for 5 consecutive days every 28 days (every month) for a total of 8 courses to low risk MDSs according to IPSS scoring system. In fact, several studies produced high rates of trilineage responses, reduces the risk of progression to acute myeloid leukemia (AML) in high-risk MDS and improves the quality of life (QoL). The use of 5-Aza in the earlier phases of MDS could reduce the proliferative advantage of MDS clone and favour the regrowth of normal hematopoiesis.

DETAILED DESCRIPTION:
5-Azacitidine(5-AZA) is the most promising drug for treatment MDSs. When administered at a dose of 75mg/m2/day subcutaneously for 7 days, every 28 days (every month), 5-Aza produces high rates of trilineage responses, reduces the risk of progression to AML in high-risk MDS and improves the QoL. The use of 5-Aza in the earlier phases of MDS could reduce the proliferative advantage of MDS clone and favour the regrowth of normal hematopoiesis. Other doses or schedules could improve its efficacy. Gene expression profile studies in MDS patients who are sensitive or resistant to 5-AZA are lacking and data coming from these studies could be useful to clarify the mechanisms of 5-azacitidine and optimize the therapy.

Objectives of the study

Primary:

* To evaluate the efficacy (hematologic response) and toxicity of 5-Aza five days monthly treatment schedule in patients with low-risk MDS (IPSS 0-INT1)

Secondary:

* To evaluate QoL by the FACT-An questionnaire
* To evaluate time to progression of MDS;
* To evaluate the gene expression profile of MDS patients sensitive or resistant to 5-AZA;
* To evaluate oncostatin M, interleukin-6 and interleukin-11 levels in the responders and non responders.

Azacitidine will be given at a dose of 75mg/sqm subcutaneous daily for 5 consecutive days every 28 days (every month) for a total of 8 courses. 5-Aza dosages will be adjusted as follows:

Patients' care and other medications

* RBC are transfused to maintain a Hb level > 90 g/L, or whenever indicated.
* Platelets are transfused if platelet count is < 20 x 109/L, or whenever indicated.
* EPO is not allowed during the trial time (8 months= 8 courses of 5-AZA therapy)
* Granulocyte or granulocyte-monocyte colony stimulating factor (G-CSF or GM-CSF) are allowed in case of severe neutropenia and/or systemic infection.
* Antibiotics and antifungals per os are given in prophylaxis if neutrophils <0.5 x 109 /L.
* Antibiotics are given i.v. in case of fever (> 38°C for > 24 h) or whenever indicated.
* Antifungals are given i.v. in case of fever persisting for more than 5 days of antibiotics i.v. or whenever indicated.
* Other experimental drugs or agents are not allowed.
* If another experimental drug or agent will be administered, the patient must discontinue the treatment with 5-AZA, and goes off-study.

Definition of Response

The response to treatment will be assessed according to IWG 2006 criteria, as reported by Cheson et al.(28) (Appendix F)

Response criteria for altering natural history of MDS:

* Complete remission (CR) Bone marrow: ≤5% myeloblasts with normal maturation of all cell lines Persistent dysplasia will be notes Peripheral blood: Hgb ≥ 11g/dl, Platelets ≥ 100 x 109/l, Neutrophils ≥ 1.0 x 109/l, Blasts 0%
* Partial remission (PR)

All CR criteria if abnormal before treatment except:

Bone marrow blasts decreased by ≥50% over pretreatment but still >5% Cellularity and morphology not relevant

* Marrow CR Bone marrow ≤ 5% myeloblasts and decrease by ≥ 50% over pretreatment Peripheral blood: if HI response, they will be noted in addition to marrow CR
* Stable disease Failure to achieve at least PR, but no evidence of progression for >8 weeks
* Failure Death during treatment or disease progression characterized by worsening of cytopenias, increase in the percentage bone marrow blasts, or progression to a more advanced MDS FAB subtype than pretreatment.
* Relapse after CR or PR

At least one of the following:

* Return to pretreatment bone marrow blast percentage
* Decrement of ≥ 50% from maximum remission/response levels in granulocytes or platelets
* Reduction in Hgb concentration by ≥ 1.5 g/dl or transfusion dependence

  * Cytogenetic Response

    1. Complete Disappearance of the chromosomal abnormality without appearance of new ones
    2. Partial At least 50% reduction of the chromosomal abnormality
  * Disease progression For patients with Less than 5% blasts: ≥50% increase in blasts to > 5% blasts 5%-10% blasts: ≥50% increase to >10% blasts 10%-20% blasts: ≥ 50% increase to > 20% blasts 20%-30% blasts: ≥50% increase to >30% blasts Any of the following At least 50% decrement from maximum remission/response in granulocytes or platelets Reduction in Hgb by ≥ 2g/dl Transfusion dependence

Survival

Endpoints:

Overall: death from any cause Event free: failure or death from any cause PFS: disease progression or death form MDS DFS: time to relapse Cause-specific death: death related to MDS

Response criteria for hematologic improvement (HI)

* Erythroid response (HI-E) (pretreatment, <11 g/dl) Hgb increase by ≥1.5 g/dl Relevant reduction on units of RBC transfusion by an absolute number of at least 4 RBC transfusions/8 weeks compared with the pretreatment transfusion number in the previous 8 weeks. Only RBC transfusions given for a Hgb of ≤ 9.0 g/dl pretreatment will count in the RBC transfusion response evaluation
* Platelet response (HI-P)(pretreatment, <100 x 109/l) Absolute increase of ≥ 30 x 109/l for patients starting with >20 x 109/l platelets Increase from < 20 x 109/l to >20 x 109/l and by at least 100%
* Neutrophil response (HI-N) (pretreatment, <1.0 x 109/l) At least 100% increase and an absolute increase > 0.5 x 109/l
* Progression or relapse after HI

  1. At least one of the following:
  2. At least 50% decrement from maximum response levels in granulocytes or platelets
  3. Reduction in Hgb by ≥ 1.5 g/dl Transfusion dependence

Quality of Life (QoL) QoL will be assessed by the FACT-An score before treatment and monthly during the study, at the end of each cycle of treatment. The FACT-An questionnaire will be performed as outpatient interviews by one trained nurse The QoL battery, according to FACT-An questionnaire, consists of items including physical, functional, emotional, social spiritual symptoms

Patient evaluation

* Physical examination (at entry and every month).
* Peripheral blood count and differential (at entry and every two weeks).
* Bone marrow biopsy (at entry; at the end of the 4th course; at the end of study-8th course).
* Bone marrow aspirate (at entry; at the end of the 4th course; at the end of study-8th course).
* Cytogenetics (at entry; at end of the 4th course; at the end of study -8th course).
* Blood biochemistry profile (at entry and every month).
* HBV, HCV, HIV (at entry).
* Gene Profile (at entry; at the end of the 4th course; at the end of study-8th course).
* Cytokines, Onc.M, IL6, IL11 (at entry; at the end of the 4th course; at the end of study-8th course).
* FACT-an (at entry; at the end of each course).

ELIGIBILITY:
Inclusion Criteria:

* Patients with low-risk (IPSS 0-INT1) MDS according to WHO classification, presenting one or more of the followings:

  * Symptomatic anemia requiring RBC transfusion supportive therapy previously unresponsive to EPO or not expected to respond to EPO
  * Thrombocytopenia requiring platelet transfusion with or without muco-cutaneous haemorrhagic syndrome
  * Persistent (> 3 months) absolute neutrophil count less then 1,5 x 109/L, with or without infections, requiring or not myeloid growth factor therapy
* ≥ 18 years old.
* Life expectancy ≥ 3 months.
* ECOG performance Status Grade 0-2.
* Serum bilirubin levels ≤ 1.5 upper limit of the normal (ULN)
* Serum GOT and GPT levels ≤ 2x UNL.
* Creatinine levels ≤ 1.5x UNL.
* Negative serum β-human chorionic gonadotropin (β-HCG) pregnancy test 24 hours prior to beginning of therapy with 5-AZA, for fertile women.
* Written informed consent.

Exclusion Criteria:

* Patients with MDS according to WHO classification with INT-2 or high IPSS risk.
* Life expectancy < 3 months.
* ECOG performance Status Grade > 2.
* Serum bilirubin levels >1.5 upper limit of the normal (ULN).
* Serum GOT and GPT levels > 2 x UNL.
* Creatinine levels >1.5 x UNL.
* Pregnancy or breast feeding.
* Insulin-dependent diabetes and uncontrolled non insulin-dependent diabetes.
* Severe cardiac or pulmonary disease incompatible with the conduction of the protocol.
* Patient with a clear indication to receive long-term anticoagulant therapy.
* Other active hematologic or solid tumors.
* Severe CNS disease.
* Malignant hepatic tumors.
* Hypersensitivity to mannitol or azacitidine.
* No written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy (hematologic response) of five days monthly 5-Aza treatment schedule in patients with low-risk MDS (IPSS 0-1). | 36 months
To evaluate the toxicity of five days monthly 5-Aza treatment schedule in patients with low-risk MDS (IPSS 0-1). | 36 months

SECONDARY OUTCOMES:
To evaluate the QoL by the FACT-An questionnaire | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof Domenico Russo, MD, Principal Investigator — Chair of Haematology, Brescia University
Locations (7):
- Italy (7):
  - University of Bologna, Bologna
  - Chair of Haematology, Bone Marrow Transplant Unit, Brescia
  - Cremona, Cremona
  - University of Genova, Genova
  - Mantova, Mantova
  - University of Siena, Siena
  - University of Udine, Udine

REFERENCES:
- [Result] Abdulhaq H, Rossetti JM. The role of azacitidine in the treatment of myelodysplastic syndromes. Expert Opin Investig Drugs. 2007 Dec;16(12):1967-75. doi: 10.1517/13543784.16.12.1967. PMID 18042004